CLINICAL TRIAL: NCT03475641
Title: Femoral Nerve Blockade in Endovenous Laser During Varicose Vein Treatment
Brief Title: Femoral Nerve Blockade in Endovenous Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Maarit Venermo, Professor in Vascular Surgery, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FEMINE
Record Dates: First submitted 2017-10-13; First posted 2018-03-23 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Pain
Keywords: pain; femoral nerve blockade; varicose vein
MeSH Terms: conditions — Pain; Varicose Veins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The current standard anesthesia (Active Comparator): Standard treatment during procedure
  Interventions: Procedure: The current standard treatment
- Femoral nerve blockade (Experimental): Femoral nerve blockade added to the standard treatment.
  Interventions: Drug: Femoral nerve blockade; Procedure: The current standard treatment

INTERVENTIONS:
Drug: Femoral nerve blockade — The femoral nerve blockade with lidocain is combined to the tumescent anesthesia.
  Arms: Femoral nerve blockade
Procedure: The current standard treatment — Tumescent anesthesia.

SUMMARY:
Varicose veins affect a majority of adult population in the western world. They decrease quality of life and may also cause venous ulcers. Therefore varicose vein treatments are justified. Currently endovenous thermal ablation is a treatment of choice for varicose veins. At the outpatient setting, however, treating both limbs at the same time may be painful to the patient especially, if simultaneous phlebectomies are performed.

The study aims to evaluate, if femoral nerve blockade can significantly decrease pain during the procedure without prolonging the stay in the hospital.

DETAILED DESCRIPTION:
Varicose veins affect a majority of adult population in the western world. They decrease quality of life and may also cause venous ulcers. Therefore varicose vein treatments are justified.

Thanks to technical advancement open surgery has been replaced By endovenous means. Currently endovenous thermal ablation is a golden standard for main trunk disease. For efficient patient and procedure flow majority of thermal ablations are performed at the outpatient setting. However, if patient is suffering from significant varicose veins, treating both legs, may be unpleasant to the patient.

Aim of the study is, whether addition of femoral nerve blockade to the tumescent anesthesia can decrease pain during the procedure without prolonging the stay in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Great saphenous vein insufficiency
* CEAP class 2-4

Exclusion Criteria:

* Neurological diseases
* Pregnancy
* CEAP 5-6
* BMI>40
* Allergy to lidocain

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Pain | Peri-procedural
  Pain analysed by Numeric Rating Scale during operation. Scale ranges from 0-10. 0 describes painless situation and 10 the worst imaginable pain ever.

SECONDARY OUTCOMES:
Pain | Pre-procedural
  Pain analysed by Numeric Rating Scale during application of anesthesia. Scale ranges from 0-10. 0 describes painless situation and 10 the worst imaginable pain ever.
Pain | 1h after the procedure
  Pain analysed by Numeric Rating Scale at 1h after the procedure. Scale ranges from 0-10. 0 describes painless situation and 10 the worst imaginable pain ever.
Motoric paresthesias of the femoral nerve | After the phlebectomies
  Ability to move knee and ankle at the end of the procedure analysed by Bromage scale. The scale measures motoric functioning of the femoral nerve: 0 = full flexion of ankle and knee possible, 1= knee flexion possible 2= ankle flexion possible, 3= impossible to move either knee or ankle
Motoric paresthesias | through study completion, an average of 1 month
  Ability to move knee and ankle one hour after the procedure analysed by Bromage scale. The scale measures motoric functioning of the femoral nerve: 0 = full flexion of ankle and knee possible, 1= knee flexion possible 2= ankle flexion possible, 3= impossible to move either knee or ankle

CONTACTS AND LOCATIONS:
Overall Officials: Anders Alback, MD,PhD, Study Chair — Head of Depratment; Karoliina H Halmesmaki, MD, PhD, Principal Investigator — Head of Venous Department
Locations (1):
- Helsinki University Hospital, Finland, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share the data is made after follow-up

REFERENCES:
- [Derived] Hurmerinta-Kurkijarvi O, Weselius EM, Halmesmaki K, Vikatmaa P, Vikatmaa L, Venermo M. Femoral nerve blockade during endovenous laser ablation of great saphenous vein decreases pain but does not affect the use of opioids during the procedure. J Vasc Surg Venous Lymphat Disord. 2023 Sep;11(5):921-927. doi: 10.1016/j.jvsv.2023.04.007. Epub 2023 May 2. PMID 37142055